CLINICAL TRIAL: NCT01000753
Title: Rare And Cutaneous Non-Hodgkin Lymphoma Registry
Brief Title: Collecting and Storing Tissue Samples From Patients With Rare or Cutaneous Non-Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANHL04B1; NCI-2009-00406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANHL04B1; CDR0000404164; ANHL04B1 (Other: Childrens Oncology Group); ANHL04B1 (Other: CTEP); U10CA098543 (NIH); UG1CA189958 (NIH)
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Adult Immunoblastic Lymphoma; Central Nervous System Non-Hodgkin Lymphoma; Childhood Immunoblastic Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3 Follicular Lymphoma; Lymphoproliferative Disorder; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Non-Hodgkin Lymphoma; Primary Cutaneous B-Cell Non-Hodgkin Lymphoma; Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoproliferative Disorders; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue, bone marrow, blood, CSF, or sera specimens

GROUPS / COHORTS (1):
- Observational (specimen collection): See Detailed Description
  Interventions: Other: Cytology Specimen Collection Procedure

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling

SUMMARY:
This research study is collecting and storing tissue samples from patients with rare or cutaneous non-Hodgkin lymphoma. Collecting and storing samples of tissue from patients with cancer to test in the laboratory may help the study of cancer in the future.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the clinical features, treatment, and outcome of patients with rare or cutaneous pediatric non-Hodgkin lymphoma (NHL).

II. To determine the pathologic and biologic features of these diseases, including molecular diagnostics and flow cytometry.

III. To establish a bank of these pathologically reviewed diseases and make specimens of blood and tissue available to qualified researchers.

IV. To determine sub-groups of these diseases that could be targeted for future biologic, pathologic, or therapeutic studies.

OUTLINE:

On study data will include presenting symptoms and signs, physical description of the tumor if it is on the skin, results of metastatic evaluation, stage (if available), blood count, markers, and the results of viral serologies. Any existing underlying conditions that could predispose to lymphoma will also be noted. Demographic and outcomes data will be stored and maintained by the COG Research Data Center. Demographic data will be linked to the specimen data in the BPC database.

The approach of this study is prospective data collection, including central pathologic review, relevant biologic studies, submission of material to the Biopathology Center (BPC) and collection of diagnostic and outcome data. Participants will be registered with a standard COG registration form for documentation of age, gender, race, date of diagnosis, initial presentation, initial work-up, and stage according to the standard staging for the specific disease, initial diagnostic procedure, and institutional diagnosis. Tissue will be sent according to guidelines in Section 4.0. Follow-up data, including relapse or progression and vital status will be reported annually for 5 years.

Patients will be followed annually for 5 years and data will be collected including vital status, evidence/absence of disease, type of treatment received, progression/relapse and whether the patient continues on study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NHL

  * Any histology, except for Burkitt or Burkitt-like, diffuse large B-cell, anaplastic large cell, or lymphoblastic lymphoma
  * Primary CNS, primary cutaneous NHL, or lymphoproliferative diseases of any histology allowed
* Pathological specimen from site not treated within the past 6 months
* Must have specimens available
* At least 6 months since prior chemotherapy irradiation to study lesion
* At least 2 weeks since prior steroids

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: PATIENTS WITH RARE OR CUTANEOUS NHL
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2005-05-30 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical features, treatment, and outcomes | Up to 5 years
Pathologic and biologic features of these diseases, including molecular diagnostics and flow cytometry | Up to 5 years
Establishment of a bank of these pathologically reviewed diseases and make specimens of blood and tissue available to qualified researchers | Up to 5 years
Sub-groups of these diseases that could be targeted for future biologic, pathologic, or therapeutic studies | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Termuhlen, Principal Investigator — Children's Oncology Group
Locations (130):
- United States (119):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, San Juan, Puerto Rico